CLINICAL TRIAL: NCT06614335
Title: An Observational Cohort Study to Explore the Clinical Outcome of Congenital Strabismmus Based on Etiology and Timing of Surgery
Acronym: strabismus
Status: Active, not recruiting | Type: Observational
Sponsor: Qiyu Bo (Other)
Responsible Party: Sponsor-Investigator, Qiyu Bo, Attending physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: CCTR-2023A02
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Congenital Esotropia
Keywords: Congenital Esotropia; Infantile Esotropia; IE; Surgical alignment rate; Stereoscopic establishment success rate
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Genetic test sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective analysis group: A retrospective analysis was performed on 220 patients who underwent IE surgery, followed up to 4 years of age, and the risk factors affecting the success rate of stereoscopic establishment were analyzed, such as strabismus, age of surgery, MRI brain features, concomitant symptoms of strabismus, etiology, refractive status, etc. The optimal timing of IE surgery and the imaging evidence related to the selection of the optimal timing were determined according to the operative orthostatic rate and the success rate of stereoscopic establishment, and the prediction model of the success rate of binocular stereoscopic establishment after surgery at different time points was constructed.
  Interventions: Other: After 6 months of observation, there was still a residual inclination of more than 15 prism degrees which needed to be corrected by a second operation
- External validation cohort of patients undergoing surgery: An externally validated retrospective analysis of 60-80 patients undergoing IE surgery was conducted to construct a prediction model for the success rate of binocular stereovision establishment after surgery at different time points.
  Interventions: Other: After 6 months of observation, there was still a residual inclination of more than 15 prism degrees which needed to be corrected by a second operation

INTERVENTIONS:
Other: After 6 months of observation, there was still a residual inclination of more than 15 prism degrees which needed to be corrected by a second operation — All IE patients enrolled were patients who had undergone corrective surgery for strabismus. Postoperative strabismus with 10 prism degrees of overcorrection or undercorrection is within the normal range. During postoperative follow-up, patients with more than 10 prism degrees of residual esotropia were treated conservally with foot orthoscopy according to their refractive status. After 6 months of observation, there were still more than 15 prism degrees of residual esotropia that needed to be corrected by a second operation. For extropia with overcorrection greater than 10 prism degrees, cross-eye training, negative mirror + prism stimulation and conservative observation and fusion training are given in the early stage, and can not be improved within 6 months, requiring a second surgical correction.

SUMMARY:
Through high-throughput sequencing and genotype/clinical phenotype/image phenotype analysis, this study will detect and find the clinical characteristics, genetic mode and gene diagnosis of children with congenital strabismus and their families, and explore the causes and pathogenesis of their diseases, so as to provide individualized treatment basis for the establishment of postoperative binocular vision in children undergoing congenital strabismus surgery. At the same time, it provides reference for the brain and intelligence development of children in the process of growth.

DETAILED DESCRIPTION:
Congenital esotropia, also known as infantile esotropia (IE), is a condition in which the eyes deviate inward at birth or within the first six months of life, with an incidence of 0.25%-0.50%. Its clinical features include a large angle of deviation with alternating gaze, the absence of binocular vision, and often accompanied by latent nystagmus, vertical disparity deviation, etc. Due to its early onset and constant nature, the damage to binocular vision function is more severe than that of other types of strabismus, and usually requires surgical correction of the eye position to improve the child's binocular vision function. However, the timing of IE surgical intervention has always been a topic of concern and controversy among doctors: some scholars believe that surgery should be performed in the early stage (within 4-6 months after birth) or the early stage (2 years before), as early surgery is beneficial to the recovery and establishment of binocular vision function in children; others argue that surgery should be performed in the late stage (2 years after birth), as if the child is too young, the preoperative examination results may not be accurate, the amount of surgery is difficult to determine, and the incidence of overcorrection and undercorrection is higher, and the improvement in visual function after surgery is not significant. Therefore, it can be seen that the earlier the surgery is performed, the higher the risk of secondary surgery; if it is too late, there is a risk of missing the opportunity to establish good stereoscopic vision. Therefore, finding the optimal surgical timing between 3 and 24 months after birth, based on the surgical alignment rate and the success rate of stereoscopic vision establishment, is an important clinical issue.

In recent years, Professor Ing M R has reported 16 cases of patients who underwent correction surgery within 6 months of birth, finding that visual quality of patients who underwent eye position correction surgery between 4-5 months after birth was not better than that of patients who underwent surgery at 6 months or older, suggesting that not all patients have the potential to establish normal binocular vision. The study reported that the occurrence of exaggerated inferior oblique muscle activity and separation of vertical deviation (DVD) after surgery can affect the recovery and establishment of binocular vision, suggesting that dysfunction of visual cortex motor processing can also affect binocular vision. Furthermore, some children with congenital esotropia were found to have hidden white matter softening lesions, suggesting that IE patients have hidden damage to brain structure. Therefore, various causes of brain structure abnormalities are important factors affecting the establishment of stereoscopic vision, and it is very necessary to use safe non-invasive imaging technology and genetic testing technology to further understand the characteristics of brain structure and function before and after surgery in IE patients, the timing of surgery, and the relationship with the establishment of binocular vision.

In recent years, increasing evidence has shown that the onset of congenital esotropia (etiology) is related to primary disorders of the visual cortex and motor processing centers in the brain of the patient: Some children with congenital esotropia were found to have hidden white matter softening lesions, cerebellar hypoplasia, or obvious decoupling trends in functional connectivity networks in brain regions, suggesting that abnormalities in brain structure and function (etiology) are closely related to eye position. More importantly, the preliminary functional MRI analysis conducted by the research team found that the longer the duration of congenital esotropia, the greater the negative impact on the child's brain structure and function network connection. After the strabismus in congenital esotropia patients was corrected by surgery, there was a widespread improvement in the functional network connection of the brain, suggesting that changes in visual experience can cause changes in human brain function and structure. Therefore, by analyzing the characteristics of brain structure and function before and after surgery in patients, it is possible to provide imaging evidence for the choice.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with congenital esotropia and treated with surgery, regardless of gender;
* Children aged 0-36 months;
* The guardian of the patient voluntarily signs the informed consent.

Exclusion Criteria:

* Esotropia found within 6 months of age due to anatomical abnormalities, extraocular muscle fibrosis, or paralysis or absence of nerves innervating the extraocular muscle;
* There are diseases or structural abnormalities affecting ocular vision development, such as congenital cataract, congenital microeyeball, congenital glaucoma, genetic or blinding eye diseases with clear genetic mutations, such as Lerber amaurosis and ocular albinism;
* Those deemed unsuitable for inclusion by the researchers.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 0-3 years of age undergoing surgery for congenital esotropia.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Orthostatic rate per operation | From enrollment to follow-up to 4 years of age
  Surgical alignment: Clinically, the standard of surgical alignment is that the postoperative eye position is less than plus or minus 10 prism degrees. Measurements are made through a prism.
Stereoscopic establishment success rate | From enrollment to follow-up to 4 years of age
  The success of stereoscopic establishment is qualitative index: yes or no. If so, further examination of fine stereoscopic acuity is performed. Titmus stereoscopic examination method was used for the examination: the examination images were composed of 3 groups: (1) Qualitative screening images of flies, which were used to quickly screen whether the subjects had stereoscopic sensation, and it was normal to perceive the float of fly wings; (2) Animal quantitative map, each row consists of 5 animal pictures, a total of 3 groups, the design parallax values are 400 ", 200 "and 100", mainly used for children under 4 years old; (3) Circle quantitative pictures, a total of 9 groups, from 800 "~ 40" divided into 9 levels of parallax. Because the above pictures are vivid, easy to use, extensive, especially suitable for children's group inspection.

SECONDARY OUTCOMES:
Secondary operation rate | From enrollment to follow-up to 4 years of age

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided